CLINICAL TRIAL: NCT01266148
Title: SCHEDULE - Scandinavian Heart Transplant Everolimus de Novo Study With Early CNI Avoidance
Brief Title: SCHEDULE - Scandinavian Heart Transplant Everolimus de Novo Study With Early Calcineurin Inhibitor (CNI) Avoidance
Acronym: SCHEDULE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001ANO02; 2009-013074-41 (EudraCT Number)
Record Dates: First submitted 2010-08-09; First posted 2010-12-24 (Estimated); Results first posted 2014-05-13 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-05

CONDITIONS: Renal Function and Chronic Allograft Vasculopathy
MeSH Terms: interventions — Cyclosporine; Mycophenolic Acid; Adrenal Cortex Hormones; Everolimus; Antilymphocyte Serum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Everolimus (Experimental): Participants started immunosuppressive regimen consisting of low dose CsA, everolimus, MMF and CS. After week 11, the participants regimen consisted of everolimus, MMF and CS.
  Interventions: Drug: Cyclosporine; Drug: Mycophenolate mofetil; Drug: Corticosteroids; Drug: Everolimus; Drug: Anti Thymocyte Globulin
- Control (Experimental): Participants received an immunosuppressive regimen consisting of CsA, MMF and CS throughout the study.
  Interventions: Drug: Cyclosporine; Drug: Mycophenolate mofetil; Drug: Corticosteroids; Drug: Anti Thymocyte Globulin

INTERVENTIONS:
Drug: Cyclosporine — Cyclosporine (CsA) control group target blood level: 150-350 ng/mL (month 1-3); 100-250 ng/mL (month 4-6); 60-200 ng/mL (month 7-12); everolimus group target blood level: 75-175 ng/mL (month 1-3)
Drug: Mycophenolate mofetil — Mycophenolate mofetil (MMF) target dose for control group: 2000-3000 mg/day everolimus group target dose: 1500-2000 mg/day and 75-175 ng/mL after week 11
Drug: Corticosteroids — Corticosteroids (CS) initiated at 0.2-0.5 mg/kg/day. Tapered to no less than 0.1 mg/kg at Month 3 for control and everolimus groups.
Drug: Everolimus — Everolimus 0.75 mg twice a day as starting dose up to a target blood level: 3-6 ng/mL (7-11 weeks) and 6-10 ng/mL for remaining of study
  Arms: Everolimus
Drug: Anti Thymocyte Globulin — Induction therapy, Anti Thymocyte Globulin (ATG): 1-2 mg/kg/day during 3-5 days for control and everolimus groups after transplant surgery and prior to randomization.

SUMMARY:
A controlled, randomized, open-label, multicenter study evaluating if early initiation of everolimus and early elimination of cyclosporine in de novo heart transplant recipients can improve long-term renal function and slow down the progression of chronic allograft vasculopathy

DETAILED DESCRIPTION:
This was a prospective, multi-center, randomized, controlled, parallel group, open label study in de novo heart transplant recipients. Patients eligibility for randomization was assessed 5 days after heart transplant.. Patients fulfilling the inclusion and exclusion criteria were randomized to one of two treatment groups: either conventional treatment with Cyclosporine A (CsA), Mycophenolate mofetil (MMF), and corticosteroids (Group A), or low-dose CsA and everolimus, reduced dose MMF, and corticosteroids (Group B). After 7 to 11 weeks, CsA was discontinued in Group B, while the standard triple-drug immunosuppressive regimen was maintained in Group A.

ELIGIBILITY:
De novo heart transplant recipients who had received induction therapy with antithomocyte globulin (ATG) were eligible for inclusion.

Recipients of multi-organ transplants or a previous transplant were excluded, as were those with a donor aged > 70 years, cold ischemia time >6 hours, patients with severe systemic infection, recipients of ABO incompatible transplants, patients with severe hypercholesterolemia (>350mg/dL) or hypertriglyceridemia (>750 mg/dL), patients with past (<5 years). In order to continue in the study after week 7-11 (period 1), patients had to complete first 7-11 weeks on randomized immunosuppression and none of the following criteria should be present: Ongoing rejection treatment or experience of one grade 3R rejection or two or more grade 2R rejections during first 7-11 weeks.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2009-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- Denmark (2):
  - Novartis Investigative Site, Århus N
  - Novartis Investigative Site, Copenhagen
- Novartis Investigative Site, Oslo, Norway
- Sweden (3):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Linköping
  - Novartis Investigative Site, Lund

REFERENCES:
- [Derived] Arora S, Andreassen AK, Karason K, Gustafsson F, Eiskjaer H, Botker HE, Radegran G, Gude E, Ioanes D, Solbu D, Dellgren G, Ueland T, Aukrust P, Gullestad L; SCHEDULE (Scandinavian Heart Transplant Everolimus De Novo Study With Early Calcineurin Inhibitors Avoidance) Investigators. Effect of Everolimus Initiation and Calcineurin Inhibitor Elimination on Cardiac Allograft Vasculopathy in De Novo Heart Transplant Recipients. Circ Heart Fail. 2018 Sep;11(9):e004050. doi: 10.1161/CIRCHEARTFAILURE.117.004050. PMID 30354362
- [Derived] Norum HM, Michelsen AE, Lekva T, Arora S, Otterdal K, Olsen MB, Kong XY, Gude E, Andreassen AK, Solbu D, Karason K, Dellgren G, Gullestad L, Aukrust P, Ueland T. Circulating delta-like Notch ligand 1 is correlated with cardiac allograft vasculopathy and suppressed in heart transplant recipients on everolimus-based immunosuppression. Am J Transplant. 2019 Apr;19(4):1050-1060. doi: 10.1111/ajt.15141. Epub 2018 Nov 5. PMID 30312541
- [Derived] Andreassen AK, Broch K, Eiskjaer H, Karason K, Gude E, Molbak D, Stueflotten W, Gullestad L; SCHEDULE (SCandinavian HEart transplant everolimus De-novo stUdy with earLy calcineurin inhibitors avoidancE) Investigators. Blood Pressure in De Novo Heart Transplant Recipients Treated With Everolimus Compared With a Cyclosporine-based Regimen: Results From the Randomized SCHEDULE Trial. Transplantation. 2019 Apr;103(4):781-788. doi: 10.1097/TP.0000000000002445. PMID 30211826
- [Derived] Nelson LM, Andreassen AK, Andersson B, Gude E, Eiskjaer H, Radegran G, Dellgren G, Gullestad L, Gustafsson F. Effect of Calcineurin Inhibitor-Free, Everolimus-Based Immunosuppressive Regimen on Albuminuria and Glomerular Filtration Rate After Heart Transplantation. Transplantation. 2017 Nov;101(11):2793-2800. doi: 10.1097/TP.0000000000001706. PMID 28230646
- [Derived] Andreassen AK, Andersson B, Gustafsson F, Eiskjaer H, Radegran G, Gude E, Jansson K, Solbu D, Karason K, Arora S, Dellgren G, Gullestad L; SCHEDULE investigators. Everolimus Initiation With Early Calcineurin Inhibitor Withdrawal in De Novo Heart Transplant Recipients: Three-Year Results From the Randomized SCHEDULE Study. Am J Transplant. 2016 Apr;16(4):1238-47. doi: 10.1111/ajt.13588. Epub 2016 Jan 28. PMID 26820618
- [Derived] Andreassen AK, Andersson B, Gustafsson F, Eiskjaer H, Radegran G, Gude E, Jansson K, Solbu D, Sigurdardottir V, Arora S, Dellgren G, Gullestad L; SCHEDULE Investigators. Everolimus initiation and early calcineurin inhibitor withdrawal in heart transplant recipients: a randomized trial. Am J Transplant. 2014 Aug;14(8):1828-38. doi: 10.1111/ajt.12809. PMID 25041227

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 115 patients (56 in the everolimus group, 59 in the control group) were randomized and received study treatment.
Pre-assignment Details: Group A (control) received treatment with Cyclosporine A (CsA), Mycophenolate mofetil (MMF), and corticosteroids.
  Group B (everolimus), received: low-dose CsA and everolimus, reduced dose MMF, and corticosteroids.
  After week 7-11, CsA was discontinued in Group B, while the standard triple-drug immunosuppressive regimen was maintained in Group A.
Period: Overall Study
Arm/Group | Everolimus | Control
Started | 56 | 59
Completed | 49 | 56
Not Completed | 7 | 3
Not completed — Adverse Event | 2 | 0
Not completed — Ongoing rejection | 1 | 0
Not completed — 2 2R rejections | 1 | 0
Not completed — Death | 2 | 3
Not completed — missing mGFR value + AE | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Everolimus | Control | Total
Number analyzed (Participants) | 56 | 59 | 115
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.02 (12.93) | 51.47 (12.36) | 51.25 (12.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 14 | 31
  Male | 39 | 45 | 84

OUTCOME MEASURES:

1. Primary Outcome: Measured Glomerular Filtration Rate (mGFR), 12 Months After Heart Transplantation
Description: Measured Glomerular Filtration Rate (mGFR) describes the flow rate of filtered fluid through the kidney. GFR is equal to the clearance rate when any solute is freely filtered and is neither reabsorbed nor secreted by the kidneys. The rate therefore measured is the quantity of the substance in the urine that originated from a calculable volume of blood. Participants' urine was used for this assessment at week 52 after heart transplant.
Time Frame: Week 52
Population: The intent to treat population includes the full analysis set patients with available data and without any major protocol deviations or criteria causing exclusion and for which data was available for analysis. Patients were analyzed according to the treatment to which they were randomized.
Measure: Mean (Standard Deviation); unit: mGFR ml/min
Arm/Group | Everolimus | Control
Number analyzed (Participants) | 51 | 56
mGFR ml/min | 79.8 (17.7) | 61.5 (19.6)

2. Secondary Outcome: Progression of Chronic Allograft Vasculopathy (CAV) Based on Maximal Intimal Thickness (MIT) From Baseline to Week 52
Description: The progression of chronic allograft vasculopathy (CAV) was assessed by intravascular ultrasound (IVUS) examinations and measured Maximal Intimal Thickness (MIT)(in mm). A major coronary epicardial artery (preferentially the left-anterior descending coronary artery) was imaged, and the MIT parameters were recorded at baseline and at week 52.
Time Frame: Baseline and week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Everolimus | Control
Number analyzed (Participants) | 46 | 48
mm
  Baseline (Week 7) | 0.52 (0.22) | 0.56 (0.24)
  Week 52 | 0.55 (0.24) | 0.65 (0.25)

3. Secondary Outcome: Progression of Chronic Allograft Vasculopathy (CAV) Based on Incidence of Chronic Allograft Vasculopathy (CAV) From Baseline to Week 52
Description: the progression of chronic allograft vasculopathy (CAV) assessed by intravascular ultrasound (IVUS) examinations, measured the incidence of CAV (in percent of patients) at baseline and at week 52. Incidence of CAV represents percent of patients having a MIT (maximal intima thickness) > 0.5 mm.
Time Frame: Baseline and week 52
Population: as for outcome 1
Measure: Number; unit: Percentage of patients
Arm/Group | Everolimus | Control
Number analyzed (Participants) | 46 | 48
Percentage of patients
  No CAV at baseline (week 7) | 43.5 | 47.9
  CAV at baseline (week 7) | 56.5 | 52.1
  No CAV at week 52 | 50 | 35.4
  CAV at week 52 | 50 | 64.6

4. Secondary Outcome: Change in Calculated Glomerular Filtration Rate From Pre-transplantation to Week 52
Description: Change in calculated glomerular filtration rate from pre-transplantation to week 52 was calculated according to the Modification of Diet in Renal Disease (MDRD) method. Measurements were taken prior to transplant (day 1), between weeks 7 to 11 and end week 52.
Time Frame: Day 1, weeks 7 to 11(baseline) and of week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mGFR mL/min
Arm/Group | Everolimus | Control
Number analyzed (Participants) | 46 | 53
mGFR mL/min
  Day 1 (n= 43, 47) | -13.0 (28.2) | -12.6 (32.6)
  Weeks 7 to 11 (n= 46, 49) | 7.4 (32.6) | -6.8 (26.2)
  Week 52 (n= 42, 53) | 27.8 (49.9) | -8.0 (28.3)

5. Secondary Outcome: Calculated Glomerular Filtration Rate From Pre-Transplantation to Week 52
Description: Calculated Glomerular Filtration Rate from pre-transplantation to week 52 was calculated according to the Modification of Diet in Renal Disease (MDRD) method. Measurements were taken prior to transplant (day 1), between weeks 7 to 11 and end of week 52.
Time Frame: Day 1, weeks 7 to 11 and of week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mGFR mL/min
Arm/Group | Everolimus | Control
Number analyzed (Participants) | 50 | 55
mGFR mL/min
  Day 1 (n= 46, 48) | 65.4 (33.8) | 66.1 (28.7)
  Weeks 7 to 11 (n=50, 51) | 84.9 (40.5) | 69.6 (19.9)
  Week 52 (n= 45, 55) | 104.5 (54.0) | 69.3 (20.4)

6. Secondary Outcome: Number of Rejections Leading to Hemodynamic Compromise
Description: Number of all rejections were recorded through the duration of the study with the intent to identify rejections leading to hemodynamic compromise.
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Number; unit: rejections
Arm/Group | Everolimus | Control
Number analyzed (Participants) | 52 | 56
rejections
  Total rejection | 185 | 128
  Treated rejection | 43 | 17
  Rejections with hemodynamic compromise | 0 | 0

7. Secondary Outcome: Occurrence of Treatment Failures up to 12 Months After Transplant
Description: Treatment failure was defined as the number of participants who died or lost their graft at any timepoint througout the duration of the study.
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Everolimus | Control
Number analyzed (Participants) | 56 | 59
participants
  Treatment failure (death) | 2 | 3
  Graff loss | 0 | 0
  Total treatment failures (graft loss + death | 2 | 3

8. Secondary Outcome: Average Level of Protenuria at Week 52
Description: Proteinuria is measured as the ratio of albumin/creatinine mg/mmol. Measurements were taken from participants urine samples.
Time Frame: 52 weeks
Population: The safety sert include all randomized participants who received at least one dose of study medication and were able to provide urine samples at week 52.
Measure: Mean (Standard Deviation); unit: mg/mmol
Arm/Group | Everolimus | Control
Number analyzed (Participants) | 52 | 56
mg/mmol | 7.2 (12.8) | 1.2 (1.4)

9. Secondary Outcome: Lipid Profile at 12 Months
Description: Total Cholesterol, LDL-Chol, HDL-Chol and TG at week 52. Measurements were taken via participants blood samples.
Time Frame: 52 weeks
Population: The safety sert include all randomized participants who received at least one dose of study medication and had blood samples taken at week 52.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Everolimus | Control
Number analyzed (Participants) | 53 | 56
mmol/L
  Total cholesterol | 5.3 (1.1) | 5.1 (1.0)
  LDL-C | 2.9 (1.0) | 2.8 (0.8)
  HDL-C | 1.6 (0.5) | 1.6 (0.5)

10. Secondary Outcome: Change in Quality of Life Assessed by SF-36 (Minnesota Living With Heart Failure Questionnaire ([MLHF)]) From Pre-transplant to Week 52 of Treatment
Description: Change in Quality of Life was assessed via the SF-36 (Minnesota Living with Heart Failure questionnaire ([MLHF)]) before transplant surgery and at week 52 of treatment. The SF-36 is a validated, self-administered questionnaire. The questionnaire, which includes 36 questions measures 8 dimensions of health: physical function, role-physical, bodily pain, general health, vitality, social function, role-emotional, and mental health. Scores can be summarized in 2 summary components assessing physical and mental health. Items in each dimension are coded, aggregated, summed, and transformed into a scale ranging from 0 (worse health) to 100 (best health).
Time Frame: Pre transplant and 52 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Everolimus | Control
Number analyzed (Participants) | 41 | 45
Units on a scale
  Physical Health pre- transplant | 30.8 (11.1) | 32.9 (8.0)
  Physical Health at week 52 | 48.8 (9.6) | 48.8 (8.3)
  Mental Health pre- transplant | 46.2 (11.8) | 38.7 (12.4)
  Mental Health at week 52 | 51.5 (12.2) | 53.9 (7.2)

11. Secondary Outcome: Change in Quality of Life - Euro Quality of Life 5D (EQ-5D)
Description: Change in Quality of Life was assessed via the EQ-5D questionnaire which consists of: EQ-5D-5L descriptive system and EQ Visual Analogue scale (EQ VAS). The EQ-5D-5L comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression). Each dimension has 5 levels (no problems, slight problems, moderate problems, severe problems, and extreme problems). The patient indicates his/her health state by checking the most appropriate statement. This decision results in a 1-digit number expressing the level selected for that dimension. The digits for 5 dimensions are combined in a 5-digit number describing the respondent's health state. The possible score is 1 to 5 where a lower number indicates improvement. The EQ VAS records the patient's self-rated health on a 20 cm vertical, visual analogue scale with endpoints labelled 'the best health you can imagine' and 'the worst health you can imagine'. The score is 0 to 100 where a higher score represents improvement.
Time Frame: Pre transplant and 52 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Everolimus | Control
Number analyzed (Participants) | 45 | 49
Units on a scale
  EQ-5D-5L pre- transplant (n=45,49) | 0.5750 (0.3387) | 0.5069 (0.3209)
  EQ-5D-5L at week 52 (n=41,44) | 0.8329 (0.2638) | 0.8367 (0.2234)
  EQ VAS pre- transplant (n=41,48) | 46.0 (24.3) | 38.9 (20.8)
  EQ VAS at week 52 (n=41,42) | 80.0 (15.0) | 79.4 (11.5)

ADVERSE EVENTS:
Groups:
- Controls: Participants received an immunosuppressive regimen consisting of CsA, MMF and CS throughout the study
Arm/Group | Controls | Everolimus
Serious Adverse Events (participants affected / at risk) | 27/59 | 27/56
Other Adverse Events (participants affected / at risk) | 53/59 | 47/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Controls (N=59) | Everolimus (N=56)
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac disorder (Cardiac disorders) | 1 | 3
Palpitations (Cardiac disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Megacolon (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Device malfunction (General disorders) | 1 | 0
Impaired healing (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 2 | 1
Pyrexia (General disorders) | 3 | 0
Bronchitis (Infections and infestations) | 1 | 1
Cytomegalovirus infection (Infections and infestations) | 3 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 1
Haemophilus infection (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 3 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 5
Sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Wound infection (Infections and infestations) | 0 | 1
Graft complication (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain stem syndrome (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 2
Psychotic disorder (Psychiatric disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pleural haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pericardial drainage (Surgical and medical procedures) | 0 | 1
Suture removal (Surgical and medical procedures) | 1 | 0
Air embolism (Vascular disorders) | 1 | 0
Femoral artery occlusion (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Controls (N=59) | Everolimus (N=56)
Anaemia (Blood and lymphatic system disorders) | 5 | 8
Leukopenia (Blood and lymphatic system disorders) | 13 | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 2
Arrhythmia (Cardiac disorders) | 9 | 6
Cardiac disorder (Cardiac disorders) | 1 | 7
Pericardial effusion (Cardiac disorders) | 2 | 4
Diarrhoea (Gastrointestinal disorders) | 2 | 10
Oedema (General disorders) | 1 | 4
Oedema peripheral (General disorders) | 10 | 12
Pyrexia (General disorders) | 1 | 3
Candidiasis (Infections and infestations) | 0 | 3
Cytomegalovirus infection (Infections and infestations) | 15 | 3
Herpes simplex (Infections and infestations) | 3 | 1
Infection (Infections and infestations) | 9 | 10
Nasopharyngitis (Infections and infestations) | 7 | 9
Pneumonia (Infections and infestations) | 1 | 4
Urinary tract infection (Infections and infestations) | 1 | 5
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 4
Gout (Metabolism and nutrition disorders) | 3 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 5
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 3
Headache (Nervous system disorders) | 1 | 3
Tremor (Nervous system disorders) | 8 | 3
Nephropathy toxic (Renal and urinary disorders) | 3 | 2
Renal failure (Renal and urinary disorders) | 3 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 | 11
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Acne (Skin and subcutaneous tissue disorders) | 1 | 6
Hirsutism (Skin and subcutaneous tissue disorders) | 4 | 0
Rash (Skin and subcutaneous tissue disorders) | 5 | 5
Hypertension (Vascular disorders) | 20 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.